CLINICAL TRIAL: NCT05631509
Title: Genetic Study of Obstructive Azoospermia
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSEC-KY-KS-2021-116
Record Dates: First submitted 2022-11-15; First posted 2022-11-30 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Genetic Disease
Keywords: CFTR; ADGRG2; Obstructive azoospermia
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA is stored at -20 degrees for 5 years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 1% of men with infertility, obstructive azoospermia (OA) may occur in congenital absence of the vas (CAVD) or idiopathic obstructive azoospermia . Many studies have shown that the pathogenic genes of OA are CFTR and ADGRG2 genes, and the inheritance mode is autosomal recessive. Although the conventional assisted reproductive technology(PESA/TESA) can help these patients have children, male patients who carry mutations of the disease-causing genes (CFTR and ADGRG2) will also pass on their mutations to the next generation, which will increase the risk of male offspring infertility. Therefore, genetic detection of CFTR and ADGRG2 genes is very necessary for CAVD patients before assisted reproduction. Genetic diagnosis plays a key role in preventing the disease to the offspring.

ELIGIBILITY:
Inclusion Criteria:

* No sperm was found after centrifugation for 15min for two or more semen tests, and the interval between two tests was at least 2 weeks.
* Blood FSH is normal;
* Hematostatin b is normal;
* Chromosome karyotype is normal or polymorphic;
* Y chromosome microdeletion did not show the deletion:(main locus);
* Biochemical fructose of seminal plasma : less than the normal value;
* PH of semen <7.2;
* Transscrotal or transrectal ultrasound: normal testicular size(as measured by B ultrasound), presence or dysplasia of vas deferens and epididymis;

Exclusion Criteria:

* B ultrasound of urinary system suggested abnormal development;
* Transscrotal or Transrectal ultrasound indicated absence of vas deferens or epididymis or seminal vesicle;
* Physical examination showed the following abnormalities: cryptorchidism, tenderness of testis and epididymis;
* The following medical history: genitourinary tract trauma or surgical history; orchitis; epididymitis; Seminal vesicle disease; mumps;
* Laboratory examination: red and white blood cell elevation of semen routine

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a non-interventional multicenter study. The cases were mainly male outpatients from the Reproductive Center of our Hospital, Shenzhen Hospital of the University of Hong Kong and Shenzhen Hospital of Traditional Chinese Medicine. A total of 300 cases were planned to be enrolled. Through inclusion criteria and exclusion criteria, appropriate patients were selected for genetic testing, including sequence of known pathogenic genes (CFTR and ADGRG2) and whole- exome sequence. If patients were found to carry mutations in CFTR, ADGRG2 or other genes, verification of family members' blood samples was required to determine the pathogenicity of mutations.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
mutation rate | through study completion, an average of 3 year
  the mutation rate of CFTR and ADGRG2

CONTACTS AND LOCATIONS:
Locations (1):
- 107 Yan Jiang Xi Road, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No